CLINICAL TRIAL: NCT00884078
Title: Exploratory RCT of Culturally Adapted Manual Assisted Problem Solving Training (C-MAP) for Self Harm in Females of South Asian Family Origin
Brief Title: Self Harm in Females of South Asian Family Origin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lancashire Care NHS Foundation Trust (Network)
Responsible Party: Louise Worrell, LCFT
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 08/H1013/6
Record Dates: First submitted 2009-02-19; First posted 2009-04-20 (Estimated); Last update posted 2009-04-20 (Estimated); Status verified 2009-04

CONDITIONS: Self Harm; Suicidal Idealtion; Hopelessness
Keywords: Self harm in south asian women; depression; suicidal ideations; problem solving training
MeSH Terms: conditions — Self-Injurious Behavior; Depression; Suicidal Ideation

ARMS (2):
- 1 (Experimental): C-MAPS (Culturally adapted manualized problem solving training) will be a brief problem focused therapy comprising of 8 sessions within three months after a self-harm episode. We will have two engagement sessions before the actual therapy. The adapted therapy/training will be delivered by therapists/trained counselors in the patient's home/GP practice depending upon patient's choice. Sessions will be offered weekly in the first month and than fortnightly and will last 50 minutes.
  Interventions: Other: Culturally adapted manualized problem solving training
- 2 Control group (No Intervention): Patients who will be randomized to the "treatment as usual" arm will receive routine care. In most cases this consists of an assessment by a casualty doctor or a junior psychiatrist in the emergency department, on the basis of which about one third patients are referred for follow up as a psychiatry outpatient, a small number are referred to addiction services, and the remainder are advised to consult their own general practitioner (Kapur 1998) this is particularly so in case of Asian females (Cooper et al, 2006). No patients are routinely referred to psychotherapy or psychology services. Participants will receive an initial assessment along with treatment as usual (TAU) as ascertained by the general practitioner or mental health professional any type of treatment apart from C-MAPS will be permitted. We will record the degree of patient adherence to standard care.

INTERVENTIONS:
Other: Culturally adapted manualized problem solving training — The areas covered by the manual include an evaluation of the self-harm attempt, crisis skills, problem solving, and basic cognitive techniques to manage emotions and negative thinking and relapse prevention strategies. The treatment will be structured around patient's current problems with the relevant sections of the manual helping the patient to deal with specific problems leading to the self-harm act. Between the sessions the manual can be used for homework tasks by the patient. We will be able to linguistically match the therapist and the participant in three most common languages spoken and understood in South Asian population i.e. Urdu, Hindi and Punjabi.
  Arms: 1

SUMMARY:
Aim of the study is to adapt and develop a culturally appropriate psychological intervention and to pilot test it's feasibility, and acceptability for the adult South Asian females presenting to general hospital emergency department following self-harm. Primary hypothesis for the study is to determine whether a brief psychological intervention compared with treatment as usual for self-harm results in decreased hopelessness and suicidal ideation. Further to this to collect necessary information on recruitment, the assessment instruments, effect size, the optimal delivery and acceptability of the intervention in preparation for a definitive RCT using repetition of self harm and cost effectiveness as the primary outcome measures.

DETAILED DESCRIPTION:
Secondary Hypothesis for the study is to compare the impact of the intervention and treatment as usual on patients' satisfaction with care, resolution of interpersonal and family problems and attributions to fully understand the mechanism of action of the intervention.

Background and Significance:

Most economically developed nations are multi-ethnic. If current demographic trends continue societies will become more ethnically diverse. UK censuses revealed that the proportion of the UK population belonging to a non-white minority ethnic group increased by 53% between 1991 and 2001, from 3 million to 4.6 million (or 7.9% of the UK population). Half of the total ethnic minority population is of south Asian family origin (UK census 2001).

Suicide, a self-directed violence, is a global public health problem. According to a recent report from the World Health Organization, world wide, suicide claimed the lives of an estimated 815,000 people in the year 2000, for an over all age-adjusted rate of 14.5 per 100,000 (WHO, 2002). In the United Kingdom, suicide is the second most common cause of death in people aged 15-24 (Hawton et al, 1998).

Prevention of suicide is now included in health policy initiatives in several countries and reduction in suicidal behavior, both fatal and non-fatal, is part of the Health for All targets of the World Health Organization (WHO, 1992). Prevention of suicide is also a priority for health services in England (Department of health, 1999a,b, 2002).

Deliberate self-poisoning is one of the commonest reasons for medical admission in the United Kingdom. (NHS Centre for R&D 1998) it is a major public health problem with over 170,000 hospital attendances per annum (Kapur et al, 1998). Health significance of attempted suicide is further underlined by the links with suicide. Of patients presenting to hospital with deliberate self-harm, up to 15% eventually kill themselves. (Nordentoft et al, 1993). It has been estimated that in the year following a suicide attempt, the risk of a repeat attempt or death by suicide may be up to 100 times greater than that seen in people who have never attempted suicide (Garland & Zigler, 1993)

Among the ethnic minority groups in UK there are reports of high rates of suicide in Asian women (Soni Raleigh et al, 1990; 1992; Neelman et al, 1996; Patel & Gaw, 1996). Previous studies from the United Kingdom have also suggested that rates of self-harm in young Asian women are higher than in the white population (Burke, 1976; Merrill & Owens, 1986; Glover et al, 1989, Husain et al, 2006). Recent hospital data in London indicate that self harm was 2.5 times more frequent among young Asian women (16-30 years) than white women of the same age and 62% of the former expressed regret that they had survived compared to 36% of the white women (Bhugra et al, 1999).

There are concerns about the acceptability of current services to ethnic minority patients (Parkman et al, 1997; Goater et al, 1999; Sashidharan, 2001). The high rate of suicide in young women of South Asian origin in the UK may be related to untreat self-harm. Of the known risk factors for suicide, the most strongly predictive of a future suicide attempt or completed suicide are hopelessness and a prior history of self harm (Brown et al, 2000).

In Manchester (MASH project) using data collected in Emergency departments over a four years period we have found a higher rate of self harm in South Asian than white European females (relative risk 1.5 times 16-24 years age group). Interpersonal conflicts within the family were the main precipitating factor, which was significantly more frequent than in white females. In spite of no differences in clinical presentation and suicidal intent there were significant differences in the Emergency departments' management of the two groups. Referral back to primary care was the most common management plan for South Asians while European whites were referred to psychiatric services for further management (Cooper et al, 2006). It is extremely important that effective treatments for deliberate self-harm patients that can be widely utilized in clinical practice be identified (Arsensman et al, 2001). We are not aware of any such intervention trials in the ethnic minorities in UK. As our population becomes increasingly diverse, tailoring practice to the area's demographics is crucial to providing effective treatment. For mental health providers in areas with large black and minority ethnic populations, it is essential to provide culturally acceptable services.

The National Service Framework (NSF) for Mental Health in UK (DoH, 1999) reaffirms the issue of inappropriate services for black and ethnic minority communities. Standard one of the NSF requires working with both individuals and communities so that disparities can be combated. The mental health services should work against social exclusion, especially with regards to people from black and minority groups. The standard seven of the NSF focuses on reduction of rates of suicide.

The NICE (National Institute of Clinical Excellence) guidelines also make recommendations for culturally sensitive services and suggest that the NHS Trusts must identify a board member to take responsibility for diversity and ethnic issues. Responsibilities must include adequacy of service provision, training on cultural difference, and monitoring service usage by ethnicity, consultation with local black and minority ethnic groups and achieving targets set in advance on a year by year basis.

The low uptake of statutory services within the South Asian community in the UK calls into question the appropriateness of the existing services. There is a need to move away from stereotypes and overgeneralizations and start from the user's frame of reference, taking account of family dynamics, belief systems and cultural constraints. This indicates the urgent need for all those concerned with the mental health services for ethnic minorities to take positive action to eradicate these barriers.

The Case for Action in Inside Outside (DOH, 2003) highlights the significantly raised risk of suicide and attempted suicide among young Asian women in the UK. Cutting the suicide rate by 20% by 2010 is a key national mental health target. Catering for the needs of this high-risk group is a vital component of meeting this target.

Under representation of ethnic minorities in mental health research: Despite the evidence for a relationship between ethnicity and increased risk for mental disorders, very little is known about providing mental health services to these groups. (Waheed et al, 2003). A new research agenda is needed to drive the development and evaluation of culturally sensitive and appropriate psychosocial interventions for ethnic minority groups. Not only studying effectiveness of these interventions but the efficiency of delivery systems as well are priorities for these special populations. (Miranda et al, 2003)

UK clinical trials are not catering for the needs of ethnic minorities (Mason 2003), unlike USA where all National Institute of health (NIH) funded research has to be sensitive to these specific needs (Sheikh 2004). This compromises their generalisability and external validity. We have ourselves carried a systematic review and have found that few studies provided information on outcomes of mental health care for ethnic minorities. In UK to date only one RCT of an educational intervention for depression has been reported (Jacob 2002). This under reporting mainly due to under-representation of ethnic minorities in health research is concerning. In fact contrary to this prevalent under investment greater resources and effort should be directed toward researching those sections of society that have the greatest capacity to benefit from such research (i.e. those at high risk and/or not currently accessing or receiving appropriate care). (Sheikh 2006)

High prevalence of suicidal ideations and depression among women of South Asian origin:

In our previous study in primary care (Husain et 1997) and in the MRC funded population-based project (Gater et al (2008)) concerning the mental health needs of people of Pakistani family origin we have demonstrated that women of Pakistani origin living in the north west of England have high rates of psychological distress and depression, 13.8% of Pakistani women from the community based sample of the 475 women reported suicidal ideations on Self Reporting Questionnaire (SRQ). This was associated with increased psychological distress (mean SRQ score of 12.3 in participants with suicidal ideas as compare to 5.23 in those who did not report suicidal thoughts). This presumably reflects the hopelessness of some South Asian women in UK.

Socio cultural determinants of deliberate self harm in women of South Asian origin:

Primary care and hospital based research in the UK has demonstrated that there are socio cultural determinants such as cultural a synchronization between women of South Asian origin and their culture of family origin characteristically in realms of overprotective home environment, differences in social norms, interpersonal conflicts with in the family, issues around personal choices like relationships and marriage as the main precipitating factors (Hicks& Bhugra 2003). Compared to match GP attenders, who had not self harmed, the Asian self-harm group was significantly less in favour of arranged marriage and was more likely to have experienced a severe life event in a close relationship (Bhugra et al, 1999b). It has been shown that younger women are not restrained by religion from being involved in self-harm as compare to older women. (Glover et al 1989). In a survey in London 180 women reported the top three causes of suicide attempts by Asian women to be 'violence by the husband' (92%), 'being trapped in an unhappy family situation' (90%), and 'depression' (90%) (Bhugra 2004).

Failure to access care as a determinant of chronic distress:

The higher rate of suicide in young women of South Asian origin (Raleigh VS, 1996) may be related to untreated self harm. A previous qualitative study has shown that young South Asian women tend to access care only at the point of desperation rather than before this crisis is reached (Chew-Graham et al 2002). There appears to be reluctance to seek early help thus prolonging the course of distress, which may be explained by a cultural attitude to mental disorders. Among South Asians, women are less likely to seek help (Fenton & Sadiq; 1993). Furthermore psychologically distressed Asian patients consulting their GP are more likely to present with a physical problem than their white counterparts, and are less likely to have their distress identified than their white counterparts (Wilson & MacCarthy1994). The literature suggests services fail to engage with ethnic minorities (Beliappa, 1991; Newham Project, 1998; Chew-Graham et al, 2001). Language problems may be a barrier to accessing appropriate treatment, although it is likely that most of the young South Asian women who self harmed were second or third generation and would be fluent in English. Low intensity of treatment and/or adverse experience of services may prevent South Asians from presenting again to hospital following subsequent self-harm episodes.

A higher proportion of South Asians (particularly women) have cited an interpersonal problem with family members as the main precipitant of the self-harm episode in our study in Manchester (Cooper et al, 2006). The psychosocial stressors which precipitate self-harm in South Asian women may be culturally influenced, but this should not exclude them from psychological help. Both problem solving therapies (Salkovskis PM et al, 1990; Hawton et al, 1998) and interpersonal forms of psychotherapy (Guthrie E et al, 1998) are of benefit in the treatment of patients who self-harm, and could potentially be of help to this group. However, work to adapt either approach, specifically to cater for the needs of South Asian women, is required. A recent systematic review of self harm concluded that while some treatments showed promise, further randomised intervention trials were required (Hawton K et al, 1998). Since most episodes of deliberate self-harm in South Asian women are precipitated by an interpersonal problem with family members there is a strong rationale for investigating the efficacy of an intervention, which addresses such issues.

Problem solving therapy has a sound theoretical basis. Consistent evidence has shown that people who attempt suicide have poor problem solving skills (Linehan, Camper, Chiles et al, 1987, Schotte & Clum, 1987; McLeavey, Day, Murray et al, 1987; Pollock & Williams, 2001). It is hypothesized that problem-solving deficits contribute to hopelessness and depression, which in turn increase the probability of suicidal ideation and intent (Schotte & Clum, 1987; D'Zurilla et al, 1998). Problem solving therapy has been found to be effective in reducing levels of depression and hopelessness in patients who have attempted suicide (Townsend et al, 2001). In addition, problem-solving therapy is a brief, cost effective, pragmatic intervention that has the potential to be widely utilized in clinical practice. Thus, the problem solving deficits seen in suicidal individuals indicate that systematic training in problem solving skills with a focus on problems precipitating the suicide attempt is likely to have a positive effect on predictors of suicidality and repetition of suicidal behavior. Thus strong rationale exists for the pilot study of problem solving therapy in order to clearly determine the acceptability of this intervention following self harm in South Asian population.

ELIGIBILITY:
Inclusion Criteria:

All females of self ascribe south Asian family origin presenting to an emergency department of the proposed study centers after an episode of self-harm.

* By self harm we mean self inflicted injury, and/or ingestion of drugs in excess of the recommended therapeutic dose, with some intention of ending one's life (Vajda and Steinbeck 2000).
* Age: 16 - 65 years
* Resident in the trial site catchment area

Exclusion Criteria:

Participants will not be excluded based on limited knowledge of English.

* Temporary resident unlikely to be available for follow up.
* ICD 10 diagnosis organic (F.0), of alcohol and drug dependence (F.1x.2) Schizophrenia (F.2) or Bipolar Affective Disorder (F.31) because these patients require a different treatment approach.
* Psychiatric admission required after deliberate self-harm.

Ages: 16 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-05; Primary Completion 2009-10 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Suicidal Ideation (Beck scale for suicidal ideation) | 6 months
Hopelessness (Beck hopelessness scale) | 6 months
Time to self-reported repetition of self harm (estimate for RCT) | 6 months

SECONDARY OUTCOMES:
Depressive symptoms assessed by Beck Depression Inventory | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nusrat Husain, Consultant Psychiatrist, Principal Investigator — LCFT
Locations (3):
- United Kingdom (3):
  - Manchester Royal Infirmary, Manchester, Greater Manchester
  - North Manchester General Hospital, Manchester, Greater Manchester
  - Royal Blackburn Hospital, Blackburn, Lancashire